CLINICAL TRIAL: NCT05849896
Title: Assistance and Evaluation of the Post-stroke Rehabilitation Process Via the Analysis of High-Density Surface EMG Signals Acquired With the WPM-SEMG-V2 Device: A Single Centre, Prospective, Feasibility Investigation in Healthy Volunteers and Post-stroke Patients
Brief Title: Clinical Relevance of the HD sEMG Signals in the Post-stroke Rehabilitation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alain Kaelin (Other)
Collaborators: University of Applied Sciences and Arts of Southern Switzerland (Other); Clinical Trial Unit Ente Ospedaliero Cantonale (Other)
Responsible Party: Sponsor-Investigator, Alain Kaelin, Principal investigator, Ente Ospedaliero Cantonale, Bellinzona
Organization: Ente Ospedaliero Cantonale, Bellinzona (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: SUPSI-SEMG-002
Record Dates: First submitted 2023-03-29; First posted 2023-05-09 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-09

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Static contractions in healthy volunteers (Experimental): Acquisition of HD SEMG signals of an upper limb muscle and a lower limb muscle while the participant executes simple static exercises.
  Interventions: Device: Acquisition of HD sEMG signals using the WPM-SEMG device
- Dynamic contractions in healthy volunteers (Experimental): Acquisition of HD SEMG signals of a leg muscle while the participant executes simple dynamic exercises.This arm will recruited recreationally active or athletic volunteers, preferably between 18 and 20 years
  Interventions: Device: Acquisition of HD sEMG signals using the WPM-SEMG device
- Static contractions in post-stroke patients (Experimental): Acquisition of HD SEMG signals of a lower limb muscle while the participant executes simple static exercises.
  Interventions: Device: Acquisition of HD sEMG signals using the WPM-SEMG device

INTERVENTIONS:
Device: Acquisition of HD sEMG signals using the WPM-SEMG device — The WPM-SEMG-V2 device will be placed over the muscle of the participant to be investigated. A reference electrode over a bone close to the muscle of investigation will be applied. A sensor combing an accelerometer, gyroscope and magnetometer integrated in the WPM-SEMG-V2 device will be also used for the acquisition of body movement measures. An additional component for trapezoidal force measurement will be used during the acquisition in static contractions to measure the force. The participant will be instructed by the investigator how to execute the static or the dynamic exercises. Visual feedback will help the subject to track the trajectory.

SUMMARY:
The goal of this clinical trial is to learn about the WPM-SEMG-V2 device (Wireless Portable and Multi-Channel, WPM) designated to acquire high-density (HD) surface electromyography (sEMG) signals in healthy volunteers and post-stroke patients. The main objectives are: 1) to technically and clinically validate the WPM-SEMG-V2 device in healthy volunteers; 2) to demonstrate the clinical relevance of the HD sEMG signals to support the process of rehabilitation of post-stroke patients. Participants will be asked to perform simple exercises using the muscles of the hand or the leg in static or dynamic contractions while wearing the WPM-SEMG-V2 device.

DETAILED DESCRIPTION:
The participant will be instructed how to execute static or the dynamic exercises while wearing the WPM-SEMG-V2 device. The WPM-SEMG-V2 device will be initially tested in a small number of healthy volunteers to evaluate the technical and clinical performance of the device in different settings (i.e., static and dynamic muscle contractions). Preliminary information gathered in the first part of the investigation may eventually guide further device modifications. The second part will capture preliminary clinical performance of the device in post-stroke patients. The main aim is to study the behaviour of the neuromuscular system in voluntary muscle activations and demonstrate the clinical relevance of the HD sEMG signals to support the process of rehabilitation of post-stroke subjects.

ELIGIBILITY:
Inclusion Criteria:

Healthy volunteers

* Written Informed Consent
* Female or male
* 18 years or older
* Ability to understand the investigation
* Willingness to complete all the investigation assessments
* Ability to perform the procedures of the investigation
* Ability to perform maximal voluntary muscle extension of the target muscle and limb

Additional inclusion criteria only for the recreationally active or athletic, healthy volunteers :

* Subjects who participated in at least 150 min of moderate activity per week over the last six months.
* between 18 and 20 years (preferably)

Post-stroke patients

* Written informed consent
* Female or male
* 18 years or older
* Have a first-time stroke
* Ability to perform maximal voluntary muscle extension of the target muscle and limb
* Preserved cognitive capacity to perform the task
* Ability to understand the investigation
* Willingness to complete all the investigation assessments
* Ability to perform the procedures of the investigation

Exclusion Criteria:

Healthy volunteers

* Any significant acute disease state
* Skin disorders/allergies at the site of contact with the investigational device
* History of skin disease
* Known hypersensitivity or allergy to component of the investigational product (e.g. metal alloys) or other materials used (e.g., abrasive gel, foam with polystyrene markers)
* Chronic use of medications or treatment

Post-stroke patients

* History of spinal cord injury or traumatic brain damage
* Serious medical illness that precludes performing the task
* Severe locomotion disorder due to other causes
* Severe neurological disease other than stroke
* Any significant acute disease state
* Skin disorders/allergies at the site of contact with the investigational device
* History of skin disease
* Known hypersensitivity or allergy to component of the investigational product (e.g. metal alloys) or other materials used (e.g., abrasive gel, foam with polystyrene markers)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-03-13 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Technical performance of the device (0 to 2) | 1 day
  Assessed during signal acquisitions in static and/or dynamic contractions in healthy volunteers by checking the following parameters:
  1. Interaction (0 or 1): when the WPM-SEMG-V2 is connected to the component for trapezoidal force measurement, both the sEMG signals and force data are recorded by the device on the device's SD card.
  2. Availability (0 or 1): all data recordings are stored separately in the SD card.
  3. Integrity of the final data (0 or 1): the recorded signals have the same duration of the recordings after post-processing of the data timestamp.
  The technical performance of the device is defined as Interaction*(availability+integrity) in static contractions.
  The technical performance of the device is the sum of the scores for availability and integrity in dynamic contractions.
Quality of the WPM-SEMG-V2 device in the acquisition of HD sEMG signals (0 to 2) | 30 days
  Assessed during signal acquisitions in static and/or dynamic contractions, both in healthy volunteers and post-stroke patients by measuring the following parameters:
  1. Signal amplitude (0 or 1): the peak-to-peak sEMG signal amplitude is within the anatomical range of few-tens of µV to 2 mV.
  2. Signal spectrum (0 or 1): the sEMG signal spectrum is within the anatomical range (sEMG power is mostly accounted for by the frequency components < 350 Hz).
  Quality of the WPM-SEMG-V2 device in the acquisition of HD sEMG signals is the sum of the scores given to signal amplitude and signal spectrum.
Correlation between the properties of populations of Motor Unit (MU) with the type of the stroke. | 30 days
  Assessed during signal acquisitions in static contractions in post-stroke patients.
  The following properties will be extracted from the MUs populations: discharge rate (pulses/seconds), recruitment threshold (percentage of the maximum voluntary force contraction), motor unit conduction velocity (meter/seconds), Muscle Fiber Conduction Velocity (meter/seconds. Type of stroke: acute or subacute.
Correlation between the properties of populations of Motor Unit (MU) with the severity of the stroke. | 30 days
  Assessed during signal acquisitions in static contractions in post-stroke patients.
  The following properties will be extracted from the MUs populations: discharge rate (pulses/seconds), recruitment threshold (percentage of the maximum voluntary force contraction), motor unit conduction velocity (meter/seconds), Muscle Fiber Conduction Velocity (meter/seconds. The severity of the stroke will be measured by the National Institutes of Health Stroke Scale (score 0-42).
Correlation between the properties of populations of Motor Unit (MU) with the location of the stroke. | 30 days
  Assessed during signal acquisitions in static contractions in post-stroke patients.
  The following properties will be extracted from the MUs populations: discharge rate (pulses/seconds), recruitment threshold (percentage of the maximum voluntary force contraction), motor unit conduction velocity (meter/seconds), Muscle Fiber Conduction Velocity (meter/seconds. The location of the stroke is obtained from MRI imaging (left hemispheric, right hemisferic, cortical, subcortical, brain stem).
Percentage of tracked MU | 30 days
  Defined as the number of tracked MU / number of detected MUs in the baseline session, among the baseline, medium term, and long term sessions. Assessed during signal acquisitions in static contractions, both in healthy volunteers and post-stroke patients

SECONDARY OUTCOMES:
Incidence of serious and non-serious adverse event, adverse device effect, device deficiency and malfunction | 30 days
  As assessed by reported adverse event.

CONTACTS AND LOCATIONS:
Overall Officials: Alain Kaelin, Prof., Study Director — Istituto di Neuroscienze Cliniche della Svizzera Italiana
Locations (1):
- Istituto di Neuroscienze Cliniche della Svizzera Italiana, Lugano, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided